CLINICAL TRIAL: NCT06750094
Title: A Randomized, Open-label Phase 3 Study of Amivantamab + FOLFIRI Versus Cetuximab/Bevacizumab + FOLFIRI in Participants With KRAS/NRAS and BRAF Wild-type Recurrent, Unresectable or Metastatic Colorectal Cancer Who Have Received Prior Chemotherapy
Brief Title: A Study of Amivantamab and FOLFIRI Versus Cetuximab/Bevacizumab and FOLFIRI in Participants With KRAS/NRAS and BRAF Wild-type Colorectal Cancer Who Have Previously Received Chemotherapy
Acronym: OrigAMI-3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 61186372COR3002; 61186372COR3002 (Other: Janssen Research & Development, LLC); 2024-513853-66-00 (Registry Identifier: EUCT number)
Expanded Access: NCT04599712 (Approved for marketing)
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms | interventions — amivantamab; Cetuximab; Bevacizumab; Fluorouracil; Leucovorin; Levoleucovorin; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Amivantamab + FOLFIRI (Experimental): Participants will receive amivantamab along with FOLFIRI (consisting of 5-fluorouracil, leucovorin calcium [folinic acid] or levoleucovorin, and irinotecan) as a chemotherapy regimen for 28-days treatment cycles and will continue to receive the treatment until radiographic disease progression or other discontinuation criteria are met.
  Interventions: Biological: Amivantamab; Drug: 5-fluorouracil; Drug: Leucovorin calcium/Levoleucovorin; Drug: Irinotecan
- Arm B: Cetuximab or Bevacizumab + FOLFIRI (Active Comparator): Participants will receive either cetuximab or bevacizumab along with FOLFIRI as a chemotherapy regimen for 28-days treatment cycles and will continue to receive the treatment until radiographic disease progression or other discontinuation criteria are met.
  Interventions: Biological: Cetuximab; Biological: Bevacizumab; Drug: 5-fluorouracil; Drug: Leucovorin calcium/Levoleucovorin; Drug: Irinotecan

INTERVENTIONS:
Biological: Amivantamab — Amivantamab will be administered.
  Other Names: JNJ-61186372
  Arms: Arm A: Amivantamab + FOLFIRI
Biological: Cetuximab — Cetuximab will be administered.
  Other Names: Erbitux
  Arms: Arm B: Cetuximab or Bevacizumab + FOLFIRI
Biological: Bevacizumab — Bevacizumab will be administered.
  Other Names: Avastin
  Arms: Arm B: Cetuximab or Bevacizumab + FOLFIRI
Drug: 5-fluorouracil — 5-fluorouracil will be administered as chemotherapy regimen.
Drug: Leucovorin calcium/Levoleucovorin — Leucovorin calcium/Levoleucovorin will be administered as chemotherapy regimen.
  Other Names: Folinic acid
Drug: Irinotecan — Irinotecan will be administered as chemotherapy regimen.

SUMMARY:
The purpose of this study is to compare how long the participants are disease-free (progression-free survival) and and the length of time until a participant dies (overall survival), when treated with amivantamab and chemotherapy with 5-fluorouracil, leucovorin calcium (folinic acid) or levoleucovorin, and irinotecan hydrochloride (FOLFIRI) versus either cetuximab or bevacizumab and FOLFIRI given to participants with Kirsten rat sarcoma viral oncogene/ neuroblastoma RAS viral oncogene homolog (KRAS/ NRAS) and v-raf murine sarcoma viral oncogene homolog B (BRAF) wild-type recurrent, unresectable or metastatic colorectal cancer who have previously received chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically confirmed adenocarcinoma of the colon or rectum. Participants must have recurrent, unresectable or metastatic disease
* Determined to have kirsten rat sarcoma viral oncogene/neuroblastoma RAS viral oncogene homolog (KRAS/NRAS), G12, G13 and v-raf murine sarcoma viral oncogene homolog B (BRAF) V600X (X represents any single amino acid change from the original amino acid) wild type status by local and/or central next-generation sequencing (NGS) testing
* Must agree to the submission of fresh or archival tumor tissue post progression from the most recent therapy, if clinically feasible
* Have measurable disease according to response evaluation criteria in solid tumors (RECIST) version (v) 1.1
* Have an eastern cooperative oncology group (ECOG) performance status (PS) of 0 or 1
* Participant must have received 1 line of systemic therapy (fluoropyrimidine-based and oxaliplatin-based) for metastatic colorectal cancer (mCRC), with documented radiographic disease progression on or after this line of therapy. Participants can receive anti-VEGF as prior line of therapy

Exclusion Criteria:

* Has medical history of (noninfectious) interstitial lung disease (ILD) /pneumonitis/pulmonary fibrosis or has current ILD/pneumonitis/pulmonary fibrosis, or where suspected ILD/pneumonitis/pulmonary fibrosis cannot be ruled out by imaging at screening
* Has known allergies, hypersensitivity, or intolerance to excipients of any of the following: amivantamab, cetuximab or bevacizumab or any component of FOLFIRI
* Has a prior or concurrent second malignancy other than the disease under study or one whose natural history or treatment is likely to interfere with any study endpoints of safety or the efficacy of the study treatment(s)
* Participant with known mismatch repair deficiency (dMMR)/ high microsatellite instability (MSI-H) status who has not received immunotherapy treatments
* Participant with known human epidermal growth factor receptor 2 (HER2)- positive/amplified tumor
* Has prior exposure to irinotecan, any agents that target epidermal growth factor receptor (EGFR) or mesenchymal epithelial transition (MET)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2029-04-13 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) as Assessed by Blinded Independent Central Review (BICR) | Up to 2 years 1 month
  PFS is defined as the time from randomization until the date of objective disease progression or death (due to any cause), whichever comes first, as assessed by BICR using response evaluation criteria in solid tumors (RECIST) version (v)1.1. Participants who have not progressed or have not died at the time of analysis will be censored at their last evaluable RECIST v1.1 assessment date.
Overall Survival (OS) | Up to 4 years 4 months
  OS is defined as the time from the date of randomization to the date of participant's death due to any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) as Assessed by BICR | Up to 4 years 4 months
  ORR is defined as the percentage of randomized participants achieving partial response (PR) or complete response (CR), as determined by BICR using RECIST v1.1 criteria.
Progression Free Survival as Assessed by Investigator | Up to 4 years 4 months
  PFS is defined as the time from randomization until the date of objective disease progression or death (due to any cause), whichever comes first, as assessed by investigator.
Objective Response Rate as Assessed by Investigator | Up to 4 years 4 months
  ORR is defined as the percentage of randomized participants achieving PR or CR, as assessed by investigator.
Duration of Response (DoR) as Assessed by BICR | Up to 4 years 4 months
  DoR is defined as time from the date of first documented response (CR or PR) until the date of documented progression or death, whichever comes first, for participants who have PR or CR as assessed by BICR.
Duration of Response as Assessed by Investigator | Up to 4 years 4 months
  DoR is defined as time from the date of first documented response (CR or PR) until the date of documented progression or death, whichever comes first, for participants who have PR or CR as assessed by investigator.
Progression Free Survival After Subsequent Therapy (PFS2) | Up to 4 years 4 months
  PFS2 is defined as the time from randomization until the date of second objective disease progression, after initiation of subsequent systemic anticancer therapy, based on investigator assessment or death, whichever comes first.
Disease Control Rate (DCR) as Assessed by BICR | Up to 4 years 4 months
  DCR is defined as the percentage of randomized participants achieving CR, PR, or stable disease (with a minimum duration of 7 weeks) as defined by BICR using RECIST v1.1.
Disease Control Rate as Assessed by Investigator | Up to 4 years 4 months
  DCR is defined as the percentage of randomized participants achieving CR, PR, or stable disease (with a minimum duration of 7 weeks) as assessed by investigator.
Time to Treatment Failure | Up to 4 years 4 months
  Time to treatment failure is defined as time from randomization to discontinuation of therapy for any reason including death, progression, toxicity, or initiation of new anticancer therapy.
Curative Resection (R0) Rate | Up to 4 years 4 months
  Curative resection (R0) rate is defined as the percentage of randomized participants who underwent curative-intent surgery where the residual tumor classification was R0.
Number of Participants with Adverse Events (AEs) by Severity | Up to 4 years 4 months
  An AE is any untoward medical occurrence in a participant administered a pharmaceutical (investigational or non investigational) product. An AE does not necessarily have a causal relationship with the treatment. Severity of AEs will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0. by using standard grades as follows: Grade 1: Mild; asymptomatic or mild symptoms; Grade 2: Moderate; minimal, local or noninvasive intervention indicated; Grade 3: Severe but not immediately life threatening; hospitalization or prolongation of hospitalization indicated; Grade 4: Life-threatening consequences; and Grade 5: Death related to AE.
Number of Participants with Abnormalities in Laboratory Values | Up to 4 years 4 months
  Participants with abnormalities in laboratory values (such as serum chemistry, hematology) will be reported.
Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score | From baseline up to 4 years 4 months
  The EORTC QLQ-C30, is a self-administered, 30-item questionnaire measuring the health-related quality of life (HRQoL) of participants with cancer. EORTC QLQ-C30 includes 5 functional scales, 3 symptom scales, a global health status / quality of life scale, and 6 single items. Responses to items 1-28 are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much." Two global health status items are rated on a 7-point numeric rating scale from 1 "Very Poor" to 7 "Excellent." Higher scores indicate greater functioning, better global health status, and more severe symptoms.
Time to Worsening in Symptoms and Functioning as Measured by EORTC QLQ-C30 | Up to 4 years 4 months
  Time to worsening in symptoms and functioning as measured by EORTC QLQ-C30 score will be reported. The EORTC QLQ-C30, is a self-administered, 30-item questionnaire measuring the health-related quality of life (HRQoL) of participants with cancer. EORTC QLQ-C30 includes 5 functional scales, 3 symptom scales, a global health status / quality of life scale, and 6 single items. Responses to items 1-28 are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much." Two global health status items are rated on a 7-point numeric rating scale from 1 "Very Poor" to 7 "Excellent." Higher scores indicate greater functioning, better global health status, and more severe symptoms.
Change From Baseline in European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C29) Score | From baseline up to 4 years 4 months
  The EORTC QLQ-CR29, is a self-administered, 29-item questionnaire measuring the HRQoL of participants with colorectal cancer. The QLQ CR29 includes items that evaluate symptoms (gastrointestinal, urinary, pain, and others) and functional areas (sexual, body image, weight, and anxiety) that are associated with colorectal cancer and its treatments. Responses are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much." All scores are linearly converted into a scale from 0 to 100. Higher scores indicate greater functioning and more severe symptoms.
Time to Worsening in Symptoms and Functioning as Measured by EORTC QLQ-C29 Score | Up to 4 years 4 months
  Time to worsening in symptoms and functioning as measured by EORTC QLQ-CR29 will be reported. EORTC QLQ-CR29, is a self-administered, 29-item questionnaire measuring the HRQoL of participants with colorectal cancer. The QLQ CR29 includes items that evaluate symptoms (gastrointestinal, urinary, pain, and others) and functional areas (sexual, body image, weight, and anxiety) that are associated with colorectal cancer and its treatments. Responses are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much." All scores are linearly converted into a scale from 0 to 100. Higher scores indicate greater functioning and more severe symptoms. Change from baseline in the EORTC QLQ-CR29 score will be reported.
Overall Side Effect Burden as Measured by European Organisation for Research and Treatment of Cancer (EORTC) Item 168 Scale Score | Up to 4 years 4 months
  EORTC item 168 is a single item used to measure the overall impact of treatment side effects. Responses are rated on a 4-point Likert response scale ranging from 1 "Not at all" to 4 "Very much. Higher scores indicates severe symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (222):
- United States (59):
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Arizona Oncology Associates PC NAHOA, Prescott, Arizona
  - St. Bernard's Medical Center, Jonesboro, Arkansas
  - CBCC Global Research, Bakersfield, California
  - Los Angeles Cancer Network, Glendale, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA, Santa Monica, California
  - Providence Medical Foundation, Santa Rosa, California
  - Torrance Memorial Physicians Network, Torrance, California
  - University of Colorado Denver Anschultz Medical Campus, Aurora, Colorado
  - Rocky Mountain Cancer Centers, Denver, Colorado
  - Eastern Connecticut Hematology & Oncology Assoc., Norwich, Connecticut
  - Florida Cancer Specialists South, Fort Myers, Florida
  - Mount Sinai Medical Center Campus, Miami Beach, Florida
  - AdventHealth Cancer Institute, Orlando, Florida
  - Florida Cancer Specialists North Region, St. Petersburg, Florida
  - Florida Cancer Specialists East, West Palm Beach, Florida
  - University Cancer And Blood Center LLC, Athens, Georgia
  - Grady Memorial Hospital, Atlanta, Georgia
  - Piedmont Cancer Institute, Atlanta, Georgia
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - Illinois CancerCare, Peoria, Illinois
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - MedStar Franklin Square Medical Center, Baltimore, Maryland
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - Cancer And Hematology Centers of Western Michigan PC, Grand Rapids, Michigan
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Washington University School Of Medicine, St Louis, Missouri
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - Astera Cancer Care, East Brunswick, New Jersey
  - Perlmutter Cancer Center at NYU Long Island, Mineola, New York
  - NYU Langone Medical Center NYU Hematology Associates, New York, New York
  - New York Cancer and Blood Specialists, Shirley, New York
  - Montefiore Einstein Comprehensive Cancer Center, The Bronx, New York
  - University Hospital of Cleveland, Cleveland, Ohio
  - Oregon Health And Science University, Portland, Oregon
  - Alliance Cancer Specialists at Main Line, Penn Wynne, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University Of Pittsburgh Medical Center UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Chattanooga, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Oncology West Texas, Abilene, Texas
  - Texas Oncology DFW, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Scott And White Memorial Hospital, Temple, Texas
  - UT Health East Texas HOPE Cancer Center, Tyler, Texas
  - Virginia Cancer Specialists, Arlington, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Providence Regional Cancer System, Lacey, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Australia (4):
  - Concord Hospital, Concord
  - Warringal Private Hospital, Heidelberg
  - Queen Elizabeth Hospital, South Woodville
  - Western Health Sunshine Hospital, St Albans
- Belgium (7):
  - Institut Jules Bordet, Anderlecht
  - UZ Antwerpen, Edegem
  - AZ Maria Middelares, Ghent
  - Jolimont, Haine Saint Paul La Louviere
  - Az Groeninge, Kortrijk
  - Universitair Ziekenhuis Leuven, Leuven
  - Centre Hospitalier Universitaire de Liege Domaine Universitaire du Sart Tilman, Liège
- Brazil (9):
  - Fundacao Pio XII, Barretos
  - Fundacao Universidade de Caxias do Sul, Caxias do Sul
  - Fundacao Doutor Amaral Carvalho, Jaú
  - Hospital Nossa Senhora da Conceicao S A, Porto Alegre
  - Hospital Santa Izabel Santa Casa de Misericordia da Bahia, Salvador
  - Fundacao Faculdade Regional De Medicina S Jose Rio Preto Hospital De Base, São José do Rio Preto
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Fundacao Antonio Prudente A C Camargo Cancer Center, São Paulo
  - Associacao Feminina de Educacao e Combate ao Cancer Hospital Santa Rita de Cassia, Vitória
- China (20):
  - Peking University First Hospital, Beijing
  - Beijing Friendship Hospital Capital Medical University, Beijing
  - Beijing Cancer Hospital, Beijing
  - The First Bethune Hospital of Jilin University, Changchun
  - Hunan Cancer hospital, Changsha
  - West China Hospital of Sichuan University, Chengdu
  - Ganzhou Cancer Hospital, Ganzhou
  - Sun Yat Sen University Cancer Center, Guangzhou
  - The Sixth Affiliated Hospital Sun Yat sen University, Guangzhou
  - Guangdong Provincial People's Hospital, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin medical university cancer hospital, Harbin
  - Huizhou Central People's Hospital, Huizhou
  - Gansu Provincial Cancer Hospital, Lanzhou
  - The First Affiliated Hospital of NanChang University, Nanchang
  - Fudan University Shanghai Cancer Center, Shanghai
  - Liaoning Cancer Hospital and Institute, Shenyang
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin
  - Hubei Cancer Hospital, Wuhan
- France (3):
  - Institut Sainte Catherine, Avignon
  - Hopital Haut Leveque, Pessac
  - CHU De Poitiers, Poitiers
- Germany (5):
  - Charite Universitatsmedizin Berlin Campus Virchow Klinikum, Berlin
  - Krankenhaus NorthWest, Frankfurt am Main
  - National Center for Tumor Diseases NCT, Heidelberg
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
  - Klinikum der Universitaet Muenchen, Munich
- Hong Kong (2):
  - Queen Mary Hospital, Hong Kong
  - Prince Of Wales Hospital, Shatin
- Hungary (3):
  - Markhot Ferenc Oktatokorhaz es Rendelointezet, Eger
  - Pecsi Tudomanyegyetem, Pécs
  - Szegedi Tudomanyegyetem, Szeged
- India (8):
  - Rajiv Gandhi Cancer Institute and Research Centre, Delhi
  - Asian Institute Of Gastroenterology, Hyderabad
  - B P Poddar Hospital and Medical research Limited, Kolkata
  - Tata Memorial Hospital, Mumbai
  - Safdarjung Hospital, New Delhi
  - Deenanath Mangeshkar Hospital and Research Centre, Pune
  - Mahamana Pandit Madan Mohan Malviya Cancer Centre, Varanasi
  - Christian medical, Vellore
- Israel (7):
  - Yitzhak Shamir Medical Center, Beer Yaakov
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta MC, Tel Aviv
- Italy (5):
  - Istituto Dei Tumori Di Milano, Milan
  - Istituto Oncologico Veneto - IRCCS, Padua
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Sanitaria Universitaria Friuli Centrale ASU FC, Udine
- Japan (10):
  - Chiba Cancer Center, Chiba
  - National Cancer Center Hospital, Chūōku
  - National Cancer Center Hospital East, Kashiwa
  - Aichi Cancer Center, Nagoya
  - National Hospital Organization Osaka National Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - Kindai University Hospital, Sakai
  - Shizuoka Cancer Center, Shizuoka
  - The University of Osaka Hospital, Suita
  - The Cancer Institute Hospital of JFCR, Tokyo
- Malaysia (6):
  - Hospital Pulau Pinang, George Town
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Umum Sarawak, Kuching
  - Institut Kanser Negara Clinical Research Center, Putrajaya
- Mexico (4):
  - Actualidad Basada En La Investigacion Del Cancer, Guadalajara
  - Centro Oncologico Personalizado Cope S De R L De C V, Mexico City
  - Health Pharma Queretaro SA de CV, Querétaro
  - COI Centro Oncologico Internacional Tijuana, Tijuana
- Netherlands (5):
  - Meander Medisch Centrum, Amersfoort
  - Antoni van Leeuwenhoek, Amsterdam
  - Radboud University Medical Center, Nijmegen
  - Erasmus MC, Rotterdam
  - ETZ TweeSteden, Tilburg
- Poland (9):
  - Bialostockie Centrum Onkologii im Marii Sklodowskiej Curie w Bialymstoku, Bialystok
  - Wojewodzki Szpital Specjalistyczny, Biała Podlaska
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im Ks B Markiewicza, Brzozów
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut BadawczyOddz w Gliwicach, Gliwice
  - Instytut Centrum Zdrowia Matki Polki, Lodz
  - SPZOZ Ministerstwa Spraw Wewnetrznych z Warminsko Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - SPZOZ Opolskie Centrum Onkologii im. Prof. Tadeusza Koszarowskiego, Opole
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
- Pan American Center for Oncology Trials LLC, San Juan, Puerto Rico
- Romania (8):
  - Centrul Medical Unirea SRL, Brasov
  - Spitalul Memorial Baneasa, Bucharest
  - Ponderas Academic Hospital, Bucharest
  - Neolife Medical Center Bucharest, Bucharest
  - Institutul Oncologic 'Prof Dr. Ion Chiricuta' Cluj-Napoca, Cluj-Napoca
  - Clinica de Oncologie Sf Nectarie, Craiova
  - Institutul Regional de Oncologie Iasi, Iași
  - Pelican Impex SRL, Oradea
- South Korea (7):
  - Kyungpook National University Chilgok Hospital, Daegu
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St Mary s Hospital, Seoul
- Spain (8):
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. Clinico Univ. de Valencia, Valencia
- Sweden (5):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Skanes universitetssjukhus, Lund
  - Sodersjukhuset, Stockholm
  - Karolinska Universitetssjukhuset, Stockholm
  - Uppsala University, Uppsala
- Taiwan (7):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- Thailand (4):
  - Ramathibodi Hospital, Bangkok
  - Siriraj Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
  - Songklanagarind hospital, Songkhla
- Turkey (Türkiye) (9):
  - Adana City Hospital, Adana
  - Gulhane Egitim ve Arastirma Hastanesi, Ankara
  - Dr Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Gazi University Hospital, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Bakirkoy Training and Research Hospital, Istanbul
  - Marmara University Pendik Training Hospital, Istanbul
  - Necmettin Erbakan University Meram Medical Faculty, Konya
  - Sakarya University Training and Research Hospital, Sakarya
- United Kingdom (7):
  - Birmingham Heartlands Hospital, Birmingham
  - Castle Hill Hospital, Hull
  - St James University Hospital, Leeds
  - St Bartholomew's Hospital, London
  - University College Hospital, London
  - Royal Marsden Hospital, London
  - Mount Vernon Cancer Centre, Northwood

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency